CLINICAL TRIAL: NCT02036827
Title: The Effect of Deep Neuromuscular Blockade on Postoperative Shoulder Tip Pain After Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Yon Hee Shim, MD, PhD, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3-2013-0210
Record Dates: First submitted 2013-12-12; First posted 2014-01-15 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Pain, Postoperative
Keywords: Pain, Postoperative; Neuromuscular Blocking Agents; Laparoscopy
MeSH Terms: conditions — Pain, Postoperative | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- moderate NMB + standard pressure (Active Comparator): Investigators will administrate rocuronium until moderate neuromuscular blockade (Train of Four >=1, Post-tetanic count>=8) is established. And pneumoperitoneum will be maintained with standard-pressure 14 mmHg.
  Interventions: Drug: Rocuronium
- deep NMB + standard pressure (Active Comparator): Investigators will administrate rocuronium until deep neuromuscular blockade (Train of Four=0, Post-tetanic count<=3) is established. And pneumoperitoneum will be maintained with standard-pressure 14 mmHg.
  Interventions: Drug: Rocuronium
- deep NMB + low pressure (Active Comparator): Investigators will administrate rocuronium until deep neuromuscular blockade (Train of Four=0, Post-tetanic count<=3) is established. And pneumoperitoneum will be maintained with standard-pressure 8 mmHg.
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium — We will administrate neuromuscular blocking agent until moderate or deep neuromuscular blockade stabilized.
  Other Names: Neurpmuscular blockade is provides vy Rocuronium Bromide

SUMMARY:
The purpose of this study was to investigate whether there is any difference in incidence of shoulder tip pain after laparoscopic cholecystectomy between the groups with moderate neuromuscular block and deep neuromuscular block.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy has become the gold standard treatment for gall bladder disease. However, 30-50% of patients suffer from shoulder tip pain, which might arise from diaphragm stretch due to pneumoperitoneum.

In the previous pilot study, working intra-abdominal space was increased in the condition of deep neuromuscular blockade. And thus investigators hypothesized that the depth of neuromuscular blockade can affect insufflation pressure and intra-abdominal volume, which result in the severity of diaphragm stretch and postoperative shoulder pain. In addition, the depth of neuromuscular blockade can alter pulmonary compliance.

ELIGIBILITY:
Inclusion Criteria:

* physical status by American society of Anesthesiology; 1 or 2 patients
* patients with benign gallbladder disease scheduled for laparoscopic cholecystectomy

Exclusion Criteria:

* patient with myasthenia gravis
* allergy to rocuronium or sugammadex
* patient with shoulder pain disease (Ex. rotator cuff tear)
* psychological disease
* patients who cannot understand Korean

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Shoulder tip pain | upto postoperative 24 hours
  The severity of shoulder tip pain will be measured in PACU and upto postoperative 6, 6-12, 12-24 hours.

SECONDARY OUTCOMES:
Postoperative pain | upto postoperative 24 hours
  The severity and the location of postoperative pain will be measured in PACU and upto postoperative 6, 6-12, 12-24 hours after operation.
Postoperative nausea and vomiting | upto postoperative 24hours
  The severity of nausea, the number of vomiting and the dose and number of administration of rescue antiemetics will be recorded.
Intraoperative hemodynamics | upto postoperative 24hours
  Heart rate and blood pressure will be measured at the completion of anesthetic induction, at the completion of carbon dioxide insufflation, at 15 minutes after carbon dioxide insufflation, at the completion of desufflation of pneumoperitoneum, and at the completion of operation.
pulmonary compliance | upto postoperative 24 hours
  Total lung compliance will be measured by the equation : CT (L/cm H2O) = change in volume/ change in pleural pressure It will be measured at the completion of anesthetic induction, at the completion of carbon dioxide insufflation, at 15 minutes after carbon dioxide insufflation, at the completion of desufflation of pneumoperitoneum, and at the completion of operation
Satisfaction of the surgeon | upto postoperative 24 hours
  Satisfaction of the surgeon will be measured by 5-scale numeric rating scale) at the completion of surgery.
Working intrabdominal space | upto postoperative 24 hours
  Working intrabdominal space will be measured by grasper (from skin to sacral promontory) at the completion of carbon dioxide insufflation.

CONTACTS AND LOCATIONS:
Overall Officials: Yon Hee Shim, MD, PhD, Study Director — Yonsei University
Locations (1):
- Gangnam severance hospital, Seoul, South Korea